CLINICAL TRIAL: NCT01395355
Title: An Integrative Intervention for Binge Eating Among Adolescent Girls
Brief Title: An Integrative Intervention for Loss of Control Eating Among Adolescent Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R34MH086922-01A2 (NIH); 1R34MH086922-01A2 (NIH)
Record Dates: First submitted 2011-06-30; First posted 2011-07-15 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Binge Eating/Loss of Control Eating
Keywords: binge eating; loss of control eating; eating in the absence of hunger; emotional eating
MeSH Terms: conditions — Bulimia; Emotional Eating

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Linking Individuals Being Emotionally Real (LIBER8) (Experimental): Participants will attend a 8-12 week, 1-2 hours long intervention comprised of cognitive behavior and dialectical behavior therapy techniques.
  Interventions: Behavioral: Linking Individuals Being Emotionally Real (LIBER8)
- Weight Management Control (Active Comparator): Participants will attend a 8-12 week, 1-2 hours long intervention comprised of behavioral weight management techniques.
  Interventions: Behavioral: Weight Management Control

INTERVENTIONS:
Behavioral: Linking Individuals Being Emotionally Real (LIBER8) — Participants will attend a 8-12 week, 1-2 hours long intervention comprised of cognitive behavior and dialectical behavior therapy techniques.
  Arms: Linking Individuals Being Emotionally Real (LIBER8)
Behavioral: Weight Management Control — Participants will attend a 8-12 week, 1-2 hours long intervention comprised of behavioral techniques.
  Arms: Weight Management Control

SUMMARY:
This study aims to develop a manualized and culturally sensitive intervention for adolescent girls targeting binge and loss of control (LOC) eating. The investigators will evaluate the feasibility and acceptability of the intervention in a controlled pilot trial. The investigators hypothesize that this intervention will serve to reduce binge and LOC eating, as well as improve psychosocial functioning as evidenced by decreased depression, anxiety, eating disorder cognitions, and impulsivity, and improved quality of life.

ELIGIBILITY:
Inclusion Criteria:

* currently meeting criteria for loss of control (LOC) eating or binge eating disorder (BED) as defined by Marcus and Kalarchian
* age 13-22
* female
* lives with parent/primary caregiver most of the time

Exclusion Criteria:

* alcohol or drug dependence in the last three months
* current suicidal intent or clinically significant self-harm behaviors reported during the assessment
* diagnosis of bulimia nervosa or anorexia nervosa in the last three months
* presence of a developmental disability or neurological impairment that would impair the individual's ability to participate in the intervention
* psychosis, including schizophrenia, or bipolar I disorder
* not fluent in English (participant and parents/primary caregivers

Ages: 13 Years to 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2011-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes in frequency of episodes of loss of control and/or binge eating from baseline to three month follow-up | 3-Month Follow-up

SECONDARY OUTCOMES:
Changes in eating disorder cognitions (e.g., eating, weight and shape concern, restrain) from baseline to three month follow-up. | 3-Month Follow-up
Changes in depressive symptoms from baseline to three month follow-up. | 3-Month Follow-up
Changes in anxiety symptoms from baseline to three month follow-up. | 3-Month Follow-up
Changes in health-related quality of life (including social, emotional, school, and physical functioning) from baseline to three month follow-up. | 3-Month Follow-up
Changes in the use of various cognitive emotion regulation strategies from baseline to three month follow-up. | 3-Month Follow-up
Changes in impulsive behaviors from baseline to three month follow-up. | 3-Month Follow-up
Changes in the frequency of eating in the absence of hunger from baseline to three month follow-up. | 3-Month Follow-up
Height and Weight | 3-Month Follow-up
Changes in the frequency of eating as a means of coping with negative emotions, such as anger, sadness and anxiety, from baseline to three month follow-up. | 3-Month Follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne E Mazzeo, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Background] Palmberg AA, Stern M, Kelly NR, Bulik C, Belgrave FZ, Trapp SK, Hofmeier SM, Mazzeo SE. Adolescent Girls and Their Mothers Talk About Experiences of Binge and Loss of Control Eating. J Child Fam Stud. 2014 Nov;23(8):1403-1416. doi: 10.1007/s10826-013-9797-z. PMID 25400491
- [Background] Mazzeo SE, Kelly NR, Stern M, Palmberg AA, Belgrave FZ, Tanofsky-Kraff M, Latzer Y, Bulik CM. LIBER8 design and methods: an integrative intervention for loss of control eating among African American and White adolescent girls. Contemp Clin Trials. 2013 Jan;34(1):174-85. doi: 10.1016/j.cct.2012.10.012. Epub 2012 Nov 9. PMID 23142669
- [Derived] Mazzeo SE, Lydecker J, Harney M, Palmberg AA, Kelly NR, Gow RW, Bean MK, Thornton LM, Tanofsky-Kraff M, Bulik CM, Latzer Y, Stern M. Development and preliminary effectiveness of an innovative treatment for binge eating in racially diverse adolescent girls. Eat Behav. 2016 Aug;22:199-205. doi: 10.1016/j.eatbeh.2016.06.014. Epub 2016 Jun 3. PMID 27299699